CLINICAL TRIAL: NCT01969162
Title: Tear Collection in Adult Volunteers
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 195263-008
Record Dates: First submitted 2013-10-21; First posted 2013-10-25 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tears
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Adult volunteers without ocular disease who have tear samples collected as per protocol. No investigational drug is administered in this study.
  Interventions: Procedure: Tear Sample Collection

INTERVENTIONS:
Procedure: Tear Sample Collection — Tear sample collection as per protocol. No investigational drug is administered in this study.

SUMMARY:
This exploratory study will collect tear samples from adult volunteers for determining and quantifying tear composition profiles. No investigational drug will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

-Adult volunteers without ocular disease.

Exclusion Criteria:

* Systemic medications that could affect eye health taken within 1 month of enrollment
* Eye infection or inflammation in either eye 3 months prior to screening
* History of herpes in either eye
* Diagnosis of dry eye or meibomian gland dysfunction
* Diagnosis of glaucoma
* Allergic conjunctivitis
* Use of rigid contact lenses within 1 year of screening
* Use of soft contact lenses within 1 week of enrollment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult volunteers without ocular disease.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Randwick, New South Wales, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Tear Lipid Composition Profile
Description: Basal (non-stimulated) tear samples were collected from one eye for lipid analysis. 13 different lipids classes were detected in individual tear samples. The concentration of each lipid class is reported in picomoles (pmole).
Time Frame: Day 1
Population: A subset of enrolled participants who had non-stimulated (basal) tear samples.
Measure: Mean (Standard Deviation); unit: pmole
Arm/Group | All Participants
Number analyzed (Participants) | 6
pmole
  Cholesterol Ester | 39.34 (6.78)
  Diacylglycerol | 0.76 (0.49)
  Free Cholesterol | 6.58 (3.11)
  Lyso- Phosphatidylcholine | 1.48 (0.71)
  Lyso- Phosphatidylethanolamine | 0.74 (0.74)
  Phosphatidylcholine | 1.43 (0.78)
  Oxygenated Phosphatidylcholine | 0.04 (0.03)
  Phosphatidylethanolamine | 0.19 (0.12)
  Phosphatidylserine | 0.21 (0.16)
  Sphingomyelin | 0.75 (0.34)
  Triacylglycerol | 2.17 (1.01)
  Wax Ester | 45.14 (5.24)
  (O-acyl)-omega-hydroxy fatty acid | 1.18 (0.60)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Screening to Day 1.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is no more than 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.